CLINICAL TRIAL: NCT03094312
Title: Evaluation of the Risk of Cognitive Deficit After Surgery of Epilepsy by Dynamic Spectral Imaging (ISD) of the Cognitive Functions in Patients Explored in StereoElectroEncephaloGraphy (SEEG)
Acronym: ISD SEEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0644; 2017-A00464-49 (Other: ID-RCB)
Record Dates: First submitted 2017-03-09; First posted 2017-03-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy
Keywords: SEEG; ISD; cognitive disorder; epilepsy surgery
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic Spectral Imaging (ISD) (Experimental): Evaluation of cognitive functions by ISD
  Interventions: Procedure: Dynamic Spectral Imaging (ISD)

INTERVENTIONS:
Procedure: Dynamic Spectral Imaging (ISD) — cerebral stimulation: dynamic spectral imaging (ISD)

SUMMARY:
Epilepsy affects between 0.5 and 0.7% of the European population. Despite the availability of numerous drug treatments, one third of patients still have seizures, which are associated with significant cognitive and social complications and excess mortality. In these patients, surgical treatment to remove the epileptogenic zone (EZ), the region of the brain responsible for seizures, is the only approach that can allow control of the disease. However, before investigating this surgery, investigations have to answer two questions: (i) what is the location and extension of the EZ and (ii) what functional risks, both motor and cognitive, would represent the resection of this Cortical region? As it is a functional surgery, it is in fact inconceivable that the surgery will result in an over-handicap. For these reasons, all candidates for surgery benefit from a complete assessment including imaging examinations, a neuropsychological assessment and a long-term video-EEG recording to record seizures. Nevertheless, in some patients, this assessment does not give us a formal answer. In these subjects, it is then necessary to carry out a second step, consisting of an invasive exploration by implantation of intracerebral electrodes during a stereoencephalography (SEEG). Due to its temporal and spatial resolution, the SEEG allows, besides the precise determination of the EZ, to carry out a functional mapping of the cortical regions likely to be included in cortectomy. Conventionally, this mapping is carried out on the basis of the cortical electrical stimulations applied to the implanted electrodes. If this approach is very robust for exploring primary functions such as motor skills or language, it cannot be used to evaluate more complex cognitive tasks such as face recognition or attention Effective cognitive treatment on a daily basis. This has led to the development in recent years, in Lyon and Grenoble, of a complementary approach to cerebral stimulation: dynamic spectral imaging (ISD). Numerous experimental paradigms have demonstrated that the realization of a cognitive task associates with the generation within the cortical regions involved in its treatment of a particular cortical activity. This activity is characterized by oscillations of the cortical rhythm in high frequencies (> 30 Hz), called gamma activities. The ISD thus consists in mapping this gamma activity during various cognitive tasks, thus making it possible to study more widely the complexity of the cognitive functions. Correlations between gamma activity and cognitive tasks have so far been exclusively performed in the non-epileptic cortex explored at the periphery of the EA during SEEG. Nevertheless, the cortical oscillatory pattern study associated with a specific cognitive task within the EZ could better anticipate complex cognitive deficits that could be generated by the resection of a cortical region.

The main objective of this project is to establish the predictive character of the gamma cortical oscillatory pattern associated with a specific cognitive task on the risk of occurrence of a cognitive disorder after surgery of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* patient adult (18-65 y/o) without legal protection measures
* Patient with a drug-resistant focal epilepsy
* Patient with a SEEG exploration as part of pre-surgical assessment of epilepsy
* patient with a consent form signed
* Intellectual capacities compatible with cognitive tasks and the signing of informed consent
* Affiliation to the social security

Exclusion Criteria:

* Pregnant women: this is already a contraindication to the realization of a SEEG study
* Subjects under 18 years of age or over 65 years of age
* Patient not suffering from EFPR, or not scheduled for SEEG
* Intellectual capacities incompatible with the cognitive tasks and / or the signature of a consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2030-01-23 (Estimated); Study Completion 2030-01-23 (Estimated)

PRIMARY OUTCOMES:
predictive character of the cortical gamma oscillatory pattern associated with a specific cognitive task on the risk of occurrence of a cognitive disorder after epilepsy surgery | 12 months post-surgery compare to preoperative assessment (SEEG)
  Relation between the presence in the epileptogenic zone of a gamma activation in at least 1 of the cognitive tasks performed during the ISD and the occurrence of a postoperative neuropsychological deficit (Wilcoxon test)

SECONDARY OUTCOMES:
database on the dynamics of large cerebral networks underlying the main cognitive functions | pre-surgical assessment (SEEG)
  Comparison of mapping of pre-surgical gamma activity with preoperative neu-ropsychological evaluation
spatio-temporal organization of these networks with that predicted by fMRI | preoperative assessment (SEEG, fMRI and cortical stimulations)
  Pre-surgical comparison of the performances for the functional cartography of gamma activity performed during SEEG, fMRI and cortical stimulation at preoperative assessment.
effect of intracerebral electrical stimulations | preoperative assessment (SEEG, fMRI and cortical stimulations)
  Pre-surgical comparison of the performances for the functional cartography of gamma activity performed during SEEG, fMRI and cortical stimulation at preoperative assessment.
macro-electrophysiological recordings | 12 months post-surgery compare to preoperative assessment (SEEG)
  The relation between the presence in the epileptogenic zone of an activation in the other frequency bands (theta, alpha, beta) in at least 1 of the cognitive tasks performed during the ISD and the occurrence of a post neuropsychological deficit
micro-electrophysiological recordings | 12 months post-surgery compare to preoperative assessment (SEEG)
  The relation between the presence in the epileptogenic zone of an activation in the other frequency bands (theta, alpha, beta) in at least 1 of the cognitive tasks performed during the ISD and the occurrence of a post neuropsychological deficit

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No